CLINICAL TRIAL: NCT05967143
Title: Observational Study to Assess Real-World Outcomes in Patients With Unresectable Liver Tumors Initiating Treatment With SIR-Spheres (Y-90 Resin Microspheres) (SIRtain Registry)
Brief Title: Observational SIR-Spheres Study for the Treatment of Unresectable Liver Tumors (SIRtain Registry)
Acronym: SIRtain
Status: Recruiting | Type: Observational
Sponsor: Sirtex Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: STX2501
Record Dates: First submitted 2023-07-07; First posted 2023-08-01 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Unresectable Hepatocellular Carcinoma (HCC); Liver Metastases From Colorectal Cancer (mCRC)
Keywords: Liver metastases from colorectal cancer (mCRC); Unresectable Hepatocellular carcinoma (HCC); SIR-Spheres microspheres; Y-90 resin microspheres; SIRT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with unresectable HCC or unresectable liver metastases from mCRC: This cohort will include patients with unresectable HCC or unresectable liver metastases from mCRC refractory to or intolerant to chemotherapy, who have been prescribed selective internal radiation therapy (SIRT) with SIR-Spheres per medical decision.
  Interventions: Device: SIRT

INTERVENTIONS:
Device: SIRT — Selective internal radiation therapy with SIR-Spheres Y90 resin microspheres.

SUMMARY:
This registry seeks to prospectively gather a large repository of comprehensive observational data reflecting routine use of SIR-Spheres in patients diagnosed with unresectable HCC or unresectable liver metastases from mCRC refractory to or intolerant to chemotherapy, in order to assess clinical response in a real-world setting and further validate the safe and appropriate use of SIR-Spheres

DETAILED DESCRIPTION:
This is a global, multi-center, prospective, observational cohort study (registry) to assess real-world outcomes in patients with unresectable HCC or unresectable liver metastases from mCRC refractory to or intolerant to chemotherapy who have been prescribed SIRT with SIR-Spheres per medical decision.

The study will be conducted through the involvement of approximately 845 patients from up to 44 sites in an estimated 10 countries.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Confirmed diagnosis of:
* Unresectable hepatocellular carcinoma (HCC) Or
* Unresectable liver metastases from colorectal cancer (mCRC) refractory to or intolerant to chemotherapy
* Identified as a candidate for SIR-Spheres treatment as deemed appropriate during the normal course of practice
* Planned to receive SIR-Spheres treatment to the liver for the first time
* Provision of signed patient informed consent

Exclusion Criteria:

* Prior radiation treatment to the liver

Caveat:

Sequential selective internal radiation therapy (SIRT) treatment is allowed

* Patients participating in any interventional clinical trial with an investigational product, device, or procedure
* Need for surrogate consent. Patients who are not able to consent on behalf of themselves are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 845 patients for whom their physicians plan to utilize SIR-Spheres in a Primary Care Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 845 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 24months from LPI
Liver PFS (LPFS) | 24months from LPI
Overall survival (OS) | 24months from LPI
Objective response rate (ORR) and liver response rate (LRR) | 24months from LPI
Duration of response (DoR) | 24months from LPI
Change scores from baseline to follow-up timepoints of the EQ-5D-5L | 24months from LPI
  The (EurolQol) EQ-5D-5L is comprised of five questions on mobility, self-care, pain, usual activities, and psychological status with 5 level answers, 5 being extreme and 1 minimum.
Change scores from baseline to follow-up timepoints of the European Organization for Research and Treatment of Cancer Quality of Life Core 30 (EORTC QLQ-C30) | 24months from LPI
  The 30 EORTC QLQ-C30 items constitute consist of 9 domains: physical function, role function, cognitive function, emotional function, social function, fatigue, pain, nausea and vomiting, and global health status. Items are answered on a scale of 1 to 4 or 1 to 7.
Change scores from baseline to follow-up timepoints of the European Organization for Research and Treatment of Cancer Quality of Life Hepatocellular Carcinoma module (EORTC QLQ-HCC18) | 24months from LPI
  The EORTC QLQ-HCC18 instrument consists of 6 symptom scales and 2 single items: that measures fatigue, body image, jaundice, nutrition, pain, fever, sexual interest and abdominal swelling. Scores are based on a 4-point Likert scale (with 1 = 'not at all' to 4 = 'very much').

SECONDARY OUTCOMES:
SAEs/SADE's rates | 24months from LPI
  Serious adverse events (SAEs)/serious adverse device effects (SADEs) rates
Subsequent hepatic procedures summarized at follow-up timepoints | 24months from LPI
  Subsequent hepatic procedures like number and type of retreatment and surgery are summarized at follow-up timepoints
Healthcare Resource Utilization summarized at follow-up timepoints | 24months from LPI
  The total HCRU of each time point specified in the protocol will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (9):
- France (3):
  - Hôpital Beaujon, Clichy, Cedex
  - Hopital Henri Mondor, Créteil, Paris
  - Hospices Civils de Lyon HCL Centre Hospitalier Lyon-Sud, Pierre-Bénite, Rhône
- Spain (3):
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (3):
  - The Christie Hospital, Manchester, Lancashire
  - Kings College Hospital, London
  - Hammersmith Hospital, London